CLINICAL TRIAL: NCT06185426
Title: Histopathological, Biochemical And Electrophysiological Evaluation Of Single Or Combined Use Of Diode Laser/Steroid Treatment On Facial Nerve Injury
Acronym: facial nerve
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Zeynep Gumrukcu, associate professor, Recep Tayyip Erdogan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RecepTayyipErdoganUni; TSA-2020-1045 (Other Grant/Funding Number: Scientific Research Projects Coordination Unit)
Record Dates: First submitted 2023-12-13; First posted 2023-12-29 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Nerve Injury; Laser Therapy; Methylprednisolone; Facial Nerve Injuries
Keywords: Facial Nerve Injury; Steroid; Low Level Laser Therapy; Nerve Recovery
MeSH Terms: conditions — Facial Nerve Injuries

STUDY DESIGN:
Intervention Model Description: Not required.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Healthy Control Group (HCG) (Placebo Comparator): Seven rats will be included randomly in this group. No surgical/medical approach will be applied.
  Interventions: Drug: Methyprednisolon and low level laser theraphy
- Damaged Control Group (DCG): (Active Comparator): Facial nerve injury will be created on the right facial nerve. No surgical/medical approach will be applied.
  Interventions: Drug: Methyprednisolon and low level laser theraphy
- Laser Group (LG) (Experimental): Facial nerve injury will be created on the right facial nerve. LLLT (Low-Intensity et al.) willl be applied 3 times a week for 4 weeks postoperatively, at 830 nm with an optical power output of 30 mW, an energy density of 4 J/cm2, an irradiation area of 0.116 cm2 and an exposure time of 16 s per spot.
  Interventions: Drug: Methyprednisolon and low level laser theraphy
- Steroid group (SG) (Experimental): Facial nerve injury will be created on the right facial nerve. Intraperitoneal methylprednisolone (1mg/kg/day) will be administered every day for 1 week postoperatively.
  Interventions: Drug: Methyprednisolon and low level laser theraphy
- Laser+Steroid Group (LSG): (Experimental): Facial nerve injury will be created on the right facial nerve. Laser and steroid treatment will be applied in combination.
  Interventions: Drug: Methyprednisolon and low level laser theraphy

INTERVENTIONS:
Drug: Methyprednisolon and low level laser theraphy — All rats will be anesthetized with ketamine hydrochloride at a dose of 50 mg/kg (i.p) (Ketalar ®, Eczacıbaşı Parke-Davis, İstanbul, Türkiye) and Xylazine HCl (Alfazyne ®, Alfasan International B.V. Woerden, Hollanda) at a dose of 10 mg/kg (intraperitoneal). A right postauricular incision will made under general anesthesia, and an external trunk of the facial nerve will be found. In the DCG and other experimental groups, the facial nerve was dissected, and it will be clamped with an average force of 150 g for about 1 minute. Afterward, the surgical area will be sutured in all rats in the DCG, L, S, and LSG groups. At the end of the 4 weeks of study, tissue samples will be taken from the facial nerve trunk in the control and experimental groups with a second surgical procedure preserved in formalin solution and sent for histopathological and biochemical examination.

SUMMARY:
The objective of the study will be to investigate the effect of low-level diode laser therapy (LLLT) and steroid on facial nerve injury. Thirty five male Wistar rat will randomly be divided into five groups: healthy control (HCG); damage control (DC); laser (LG); steroid (SG); and combined laser and steroid group (LSG). Right facial nerve electromyography (EMG) data will record after facial nerve damage done and before sacrification at 4th week.The results will be evaluated histopathologically, electrophysiologically and biochemically.

DETAILED DESCRIPTION:
The animals will be randomly divided into two control groups, a healthy control group and a damaged control group, and three experimental groups; 7 rats were assigned to each group as follows;

1. Healthy Control Group (HCG): Seven rats will be included randomly in this group. No surgical/medical approach will be applied. EMG measurements will betaken over the right facial nerve.
2. Damaged Control Group (DCG): Facial nerve injury will be created on the right facial nerve. No surgical/medical approach will be applied. EMG measurements will be taken over the right facial nerve after the injury and after the four weeks of treatment.
3. Laser Group (LG): Facial nerve injury will be created on the right facial nerve. LLLT (Low-Intensity et al.) will be applied 3 times a week for 4 weeks postoperatively, at 830 nm with an optical power output of 30 mW, an energy density of 4 J/cm2, an irradiation area of 0.116 cm2 and an exposure time of 16 s per spot. EMG measurements will be taken over the right facial nerve after the injury and after the four weeks of treatment.
4. Steroid group (SG): Facial nerve injury will be created on the right facial nerve. Intraperitoneal methylprednisolone (1mg/kg/day) will be administered every day for 1 week postoperatively. EMG measurements will be taken over the right facial nerve after the injury and after the four weeks of treatment.
5. Laser+Steroid Group (LSG): Facial nerve injury will be created on the right facial nerve. Laser and steroid treatment will be applied in combination. EMG measurements will be taken over the right facial nerve after the injury and after the four weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

-Thirty-five male Sprague-Dawley rats weighing 200-300 g will be included the study

Exclusion Criteria:

-Rats that are older than 6 months and are not healthy and have impaired facial motor functions will be excluded from the study.

Ages: 4 Months to 6 Months | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Electromyographic Analysis | 1 month
  Measuring the amplitude and latency of the action potential occurring in the nerve with electromyography(On facial nerve)

SECONDARY OUTCOMES:
Biochemical Analysis | 1 month
  Determination of MDA and GSH levels in blood samples taken

CONTACTS AND LOCATIONS:
Overall Officials: zeynep gümrükçü, Associate Professor, Study Director — RTEU
Locations (1):
- RTEU Faculty of Dentistry, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No